CLINICAL TRIAL: NCT06101654
Title: Accuracy of the Evie Ring Pulse Oximeter in Profound Hypoxia
Brief Title: Accuracy of Evie Ring Pulse Oximeter in Profound Hypoxia
Status: Completed | Type: Observational
Sponsor: Movano Health (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: MOVA05
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Adult Volunteers: Minimum of ten (10) subjects meeting the eligibility criteria.
  Interventions: Device: Pulse oximeter

INTERVENTIONS:
Device: Pulse oximeter — Devices (4) were placed on the finger and the fingertip of both index fingers. Blood samples were taken at each stable level of oxygenation.

SUMMARY:
The goal of this study was to evaluate the accuracy of pulse oximeters over the range of 70-100% per ISO 80601-2-61:2019. Four devices were placed on each subject with two on each index finger at the base and two on each index finger at the fingertip. SpO2 measurements from these devices were compared to sampling of arterial blood during brief stable oxygen desaturation in healthy volunteers to evaluate the claimed range.

DETAILED DESCRIPTION:
The study is an open enrollment, single-center, single blinded design using the investigational ring compared to arterial blood gas measurements (SaO2) and to two commercially available hospital grade reference pulse oximeters (Massimo Radical-7 and Nellcor N-595). To be included in the study, subjects had to meet all the inclusion criteria and not meet any of the exclusion criteria and to sign the written consent. Demographic data were obtained.

The investigational (4/subject) and reference devices were placed. A radial arterial cannula was placed in either the left or right wrist of each subject for arterial blood sampling and blood pressure monitoring. Each subject had two control blood samples taken at the beginning of each experiment, while breathing room air. Hands with test devices and reference pulse oximeters were maintained motionless on arm boards throughout the test. Hypoxemia was then induced to different and stable levels of oxyhemoglobin saturation (between 70-100%) by having subjects breathe mixtures of nitrogen, air, and carbon dioxide. The mixture of gases was controlled by the study physician by adjusting gas flows according to breath-by-breath estimates of oxygen saturation calculated from end-tidal partial pressure of oxygen (PO2) and partial pressure of carbon dioxide (PCO2). Each plateau level of oxyhemoglobin saturation was maintained for at least 30 seconds or until readings were stable. Two arterial blood samples were then obtained, approximately 30 seconds apart. Each stable plateau was maintained for at least 60 seconds with SpO2 fluctuating by less than 2-3%. All investigational, control, and reference data were recorded.

ELIGIBILITY:
Inclusion Criteria:

Subject is in good general health with no evidence of any medical problems. Subject is fluent in both written and spoken English. Subject provided written informed consent and is willing to comply with the study procedures.

Subject is willing to have their skin color assessed.

Exclusion Criteria:

Subject is obese with a BMI over 30. Subject has a known history of heart disease, lung disease, kidney or liver disease.

Subject has asthma, sleep apnea, or uses a CPAP. Subject has diabetes. Subject has a clotting disorder, anemia, or in the opinion of the investigator, they would be unsuitable for participation.

Subject has any other serious system illness. Subject is a current smoker. Subject has any injury, deformity, or abnormality at the sensor sites that, in the opinion of the investigator, would interfere with the sensors working correctly.

Subject has a history of fainting or vasovagal response. Subject has a sensitivity to local anesthesia. Subject has Raynaud's disease. Subject has unacceptable collateral circulation based on an exam by the investigator.

Subject is pregnant, lactating, or trying to get pregnant. Subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with the study procedures.

Subject has any other condition, which in the opinion of the investigator, would make them unsuitable for the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult participants 18 to 49 years old, of which 2 or 15% of the subject pool is darkly pigmented.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
RMSE compared to arterial blood SaO2 | 2 days
  Root Mean Squared Error between Movano Ring SpO2 measurement and the arterial blood SaO2 calibrated using arterial blood gas.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, MD, PhD, Principal Investigator — University of California at San Francisco (UCSF)
Locations (1):
- Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No